CLINICAL TRIAL: NCT01967875
Title: A Prospective, Multi-Center, Randomized Control Phase 2 Trial of Optimizing Platinum-Based Chemotherapy Based on ERCC1 Expression as First-Line Treatment in Patients With Locally Advanced or Metastatic Gastric Cancer
Brief Title: A Phase 2 Trial of Optimizing Platinum-Based Chemotherapy Based on ERCC1 Expression as First-Line Treatment in Patients With Locally Advanced or Metastatic Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, MD.,PhD, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1301
Record Dates: First submitted 2013-10-15; First posted 2013-10-23 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Stomach Neoplasms
Keywords: Gastric Cancer; ERCC1; Platinum; Chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- H-A: ERCC1 High Expression Group A (Active Comparator): XP：Capecitabine+Cisplatin
  Interventions: Drug: Capecitabine+Cisplatin
- H-B: ERCC1 High Expression Group B (Experimental): DX：Docetaxel+Capecitabine
  Interventions: Drug: Docetaxel+Capecitabine
- L: ERCC1 Low Expression Group (Active Comparator): XP：Capecitabine+Cisplatin
  Interventions: Drug: Capecitabine+Cisplatin

INTERVENTIONS:
Drug: Capecitabine+Cisplatin — Cisplatin 75mg/m2, d1; Capecitabine 1700-2000mg/m2/day on days1-14 every 21 days, 6 cycles.Capecitabine is to be continued until disease progression or intolerable toxicity.
  Other Names: Xeloda
  Arms: H-A: ERCC1 High Expression Group A; L: ERCC1 Low Expression Group
Drug: Docetaxel+Capecitabine — Docetaxel 75mg/m2, d1; Capecitabine 1700-2000mg/m2/day on days1-14 every 21 days, 6 cycles. Capecitabine is to be continued until disease progression or intolerable toxicity.
  Other Names: Docetaxel for injection; Xeloda
  Arms: H-B: ERCC1 High Expression Group B

SUMMARY:
The purpose of this study is to determine whether ERCC1(excision repair cross-complementation 1 ) expression has effects on platinum-based chemotherapy for patients with locally advanced or metastatic gastric cancer, and to explore if ERCC1 can act as a biological predictor for the individual therapy of gastric cancer

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized control clinical trial, aimed to demonstrate if ERCC1 expression could predict the efficacy of platinum-based chemotherapy in patients with locally advanced or metastatic gastric cancer. A total of 180 patients are planned to be enrolled into the study. ERCC1 protein expression in paraffin-embedding tumor tissue is examined by immunohistochemistry (IHC). Patients with low ERCC1 expression (group L) will be treated with XP regimen. Patients with high ERCC1 expression will be randomized into group H-A or group H-B, and be treated with XP or DX regimen, respectively. The primary end point is progression free survival (PFS), and the secondary end points include the median overall survival, objective response rate (ORR),disease control rate(DCR), duration of response, safety(number and degree of adverse events), and the quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

* 18y≤Age≤65y, male or female
* KPS≥70
* Histologically confirmed adenocarcinoma of the stomach or gastro-oesophageal junction with inoperable locally advanced or recurrent and/or metastatic disease
* At least one measurable lesion, according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), assessed using imaging techniques (CT or MRI)
* No prior anti-tumor treatment or an interval of at least 6 months from the last adjuvant chemotherapy, and an interval of at least 4 weeks from the last radical radiation therapy
* No major organ disorder, with normal liver, kidney and heart function
* Laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count ≥1.5×109/L, platelet count ≥100×109/L, creatinine clearance rate (CCr) ≥60ml/min, total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), blood glucose ≤11.1 mmol/L
* Life expectancy of at least 12 weeks
* Signed informed consent
* For women with child bearing potential, a negative serum or urine pregnancy test result should be obtained before enrollment

Exclusion Criteria:

* Progression from prior palliative treatment with capecitabine- or docetaxel-based regimen
* Serious uncontrolled systemic illness or medical condition: congestive heart failure, unstable angina, history of documented myocardial infarction within 6 months, uncontrolled hypertension and high risk uncontrollable arrhythmias; Obvious neurological or mental abnormalities including mental disorder, epileptic dementia, which affect compliance; Uncontrolled acute infections; Uncontrolled peptic ulcer, diabetes or other contraindication for corticosteroid therapy
* Inability to take or absorb oral medicine
* Concurrent administration of any other investigational drug, or have been enrolled in other clinical trial with investigational drug treatment within the 30 days of start of study treatment
* Presence of neuropathy ≥grade 1 according to NCI-CTCAE V4.0
* Hypersensitivity or known or suspicious allergic to any of the study drugs
* Pregnant or lactated women
* Unsuitable for the study or other chemotherapy determined by investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
Objective Response Rate(ORR),Including Complete Response(CR) and Partial Response(PR) | 2 years
Disease Control Rate(DCR), Including Complete Response(CR) , Partial Response(PR) and Stable Disease(SD) | 2 years
Duration of Response | 2 years
Safety(number and degree of adverse events) | 2 years
Quality of Life(QOL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, MD., PhD, Principal Investigator — China Medical University, China; Xiujuan Qu, MD.,PhD., Principal Investigator — China Medical University, China
Locations (7):
- China (7):
  - The Fourth Hospital of Anshan, Anshan, Liaoning
  - The First Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of Liaoning Medical University, Jinzhou, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Tumor Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning